CLINICAL TRIAL: NCT02483182
Title: A Phase II, Randomized, Double-Blind, Parallel Group, Acyclovir-Controlled Study to Evaluate ZEP-3 Ointment for the Treatment of Cold Sores (Herpes Labialis).
Brief Title: Safety, Tolerability and Therapeutic Efficacy of Topical ZEP-3 Ointment (1.0%) for the Treatment of Cold Sores
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shulov Innovate for Science Ltd. 2012 (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZEP - 002 - IL
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2018-04

CONDITIONS: Herpes Labialis
Keywords: Herpes labialis, Cold sores, ZEP-3 ointment
MeSH Terms: conditions — Herpes Labialis | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZEP-3 ointment 1.0% (Experimental): Topical administration
  Interventions: Drug: ZEP-3 ointment 1.0%
- Acyclovir cream 5% (Active Comparator): Topical administration
  Interventions: Drug: Acyclovir cream 5%

INTERVENTIONS:
Drug: ZEP-3 ointment 1.0%
  Arms: ZEP-3 ointment 1.0%
Drug: Acyclovir cream 5%
  Other Names: Zovirax
  Arms: Acyclovir cream 5%

SUMMARY:
This is a phase II, prospective, randomized, double-blind, parallel group, acyclovir-controlled clinical study to evaluate the safety, tolerability and preliminary therapeutic efficacy of ZEP-3 ointment 1.0% for the treatment of cold sores (Herpes labialis), following five consecutive treatment days with five times daily topical administration.

DETAILED DESCRIPTION:
The primary endpoint of this study are:

* "Time to healing" - Clinician-assessed duration in days of herpes labialis episode.
* Patient-assessed duration and intensity of pain by Visual Analog Scale (VAS).
* Safety and tolerability following five consecutive treatment days with five times daily topical administration.

The secondary endpoints of this study are:

* Proportion of subjects with non - ulcerative herpes lesion.
* Time for herpes labialis recurrences

Subject safety will be assessed following treatment by ZEP-3 ointment 1.0% or acyclovir cream 5% treatment, using measurements of the following variables:

* Physical examination,
* Vital Signs (HR, BP, Body temperature),
* Adverse events recording and
* Concomitant medications

ELIGIBILITY:
Inclusion Criteria:

Prior to enrollment in this study, candidates must meet ALL of the following inclusion criteria:

1. Patients suffering from recurrent Herpes labialis with history of at least 3 cold sores recurrences during the previous 12 months.
2. Participants, either male or female are between 18 and 75 years of age.
3. Patients arrive at the clinic with any symptom of an acute Herpes labialis episode.

   Or, patients arrive at the clinic within 48 hours of treatment initiation for a recurrent Herpes labialis episode.
4. Patients with previous Herpes labialis episode must be healed for at least 14 days before baseline visit
5. Patients with no history of reaction to topical products.
6. Female subjects of childbearing potential must have a negative pregnancy test at screening and agree to use a proper contraceptive method during the study.
7. Participant understands the nature of the procedure and is willing and able to comply with all requirement of the protocol.
8. Patient is willing and able to provide written informed consent prior to any study procedure.

Exclusion Criteria:

1. Subject has abnormal skin conditions or significant facial hair at or near the investigational area
2. Subject has any body piercing in or around the area ordinarily affected by cold sores.
3. Subjects with a history of cardiac abnormalities.
4. Subject has a recent history of renal dysfunction or serious hepatic disease
5. Subject has an active malignancy or immunodeficient disease
6. Subject who is unwilling to stop using topical medical, OTC, cosmetics or facial skin care products in or around the oral area during the study period.
7. Subject requires chronic use of immunomodifying drugs or topical steroids on or near the face.
8. Subject requires chronic use of anti-viral medication.
9. Subject requires chronic use of analgesics, pain medication or non-steroidal anti inflammatory agents (NSAIDs).
10. History of allergic or adverse response to acyclovir, or any related anti-viral drug.
11. Subject has had an infection with HSV-1 isolates know to be resistant to acyclovir, valacyclovir, famciclovir, or ganciclovir.
12. Subject has had a herpes vaccine.
13. Females during pregnancy, lactation or breastfeeding.
14. Subject has a history of alcoholism or drug abuse within the preceding 12 months.
15. Subject is currently enrolled in another clinical trial involving the use of a drug and/or a device.
16. Any history which, in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk.
17. Subjects with immune deficiency conditions including acquired immune deficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06-24 (Actual); Study Completion 2018-06-24 (Actual)

PRIMARY OUTCOMES:
Clinician-assessed "Time to healing" | Up to 14 days

SECONDARY OUTCOMES:
Time for Herpes labialis recurrences | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shemer Avner, Prof., M.D., Principal Investigator — Dermatology out-patients clinic, Lev Hayasmin - Medical center, Natanya, ISRAEL
Locations (1):
- Dermatology out-patients clinic, Lev Hayasmin MC, Netanya, Israel